CLINICAL TRIAL: NCT00404404
Title: Phase II Trial of Abraxane Administered on a Weekly Schedule in Combination With Bevacizumab in Metastatic Breast Cancer
Brief Title: ABI-007 and Bevacizumab in Treating Women With Recurrent or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Premiere Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000515534; PREMIERE-AVF3678s; PREMIERE-20061500; GENENTECH-PREMIERE-AVF3678s; ABRAXIS-PREMIERE-AVF3678s
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Taxes

INTERVENTIONS:
Biological: bevacizumab
Drug: paclitaxel albumin-stabilized nanoparticle formulation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ABI-007, work in different ways stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving ABI-007 together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II is studying how well giving ABI-007 together with bevacizumab works in treating women with recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity of paclitaxel albumin-stabilized nanoparticle formulation (ABI-007; Abraxane^®) and bevacizumab, in terms of progression-free survival and response rate, in women with recurrent or metastatic breast cancer.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Determine the feasibility of this regimen in these patients.

OUTLINE: This is an open-label, pilot study.

Patients receive paclitaxel albumin-stabilized nanoparticle formulation (ABI-007; Abraxane^®) IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive breast cancer
* Recurrent or metastatic disease OR locally recurrent disease not amenable to resection with curative intent
* Measurable or nonmeasurable disease
* No CNS metastases by CT scan or MRI
* No HER2-neu-positive tumors
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count > 100,000/mm³
* Creatinine < 2.0 mg/dL
* Bilirubin normal
* AST ≤ 2 times upper limit of normal (ULN) (5 times ULN if there is known liver involvement)
* Urine protein:creatinine ratio < 1.0 OR proteinuria < 2+ by urine dipstick OR ≤ 1 g protein on 24-hour urine collection
* No peripheral neuropathy > grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancies within the past 5 years except carcinoma in situ of the cervix, melanoma in situ, or basal cell carcinoma of the skin
* No inadequately controlled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg and/or diastolic BP > 100 mm Hg on antihypertensive medications
* No prior hypertensive crisis or hypertensive encephalopathy
* No New York Heart Association class II-IV congestive heart failure
* No myocardial infarction or unstable angina within the past 6 months
* No stroke or transient ischemic attack within the past 6 months
* No significant vascular disease (e.g., aortic aneurysm or aortic dissection)
* No symptomatic peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious, nonhealing wound, ulcer, or bone fracture
* No known hypersensitivity to any component of bevacizumab

PRIOR CONCURRENT THERAPY:

* No prior paclitaxel albumin-stabilized nanoparticle formulation (ABI-007; Abraxane^®) or bevacizumab
* No prior chemotherapy for metastatic disease
* Prior hormonal therapy for metastatic disease allowed
* At least 4 weeks since any prior therapy for cancer

  * More than 12 months since prior adjuvant chemotherapy, including use of a taxane
* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior core biopsy or minor surgery (excluding placement of a vascular access device)
* No concurrent major surgery
* No other concurrent therapy for breast cancer
* Concurrent bisphosphonates allowed if there is bone involvement
* No concurrent prophylactic granulocyte colony-stimulating factors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Progression-free survival as measured by RECIST criteria at 1 and 2 years

SECONDARY OUTCOMES:
Response rate measured every 3 courses during treatment
Overall survival
Time to progression
Disease-free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Chap, MD, Principal Investigator — Premiere Oncology
Locations (1):
- Premiere Oncology, Santa Monica, California, United States